CLINICAL TRIAL: NCT05634135
Title: The Difference and Prognostic Significance of Lung Ventilation and Perfusion in Different Phenotypes of Chronic Critical Illness With Prolonged Mechanical Ventilation
Brief Title: Lung Ventilation and Perfusion in Different Phenotypes of Chronic Critical Illness With Prolonged Mechanical Ventilation
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202112183RIND
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-09

CONDITIONS: Prolonged Mechanical Ventilation
Keywords: Ventilation; mechanical ventilation; weaning; oxygen uptake
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project will conduct a series of analysis of physiological and clinical data on tracheostomy patients who receive prolonged mechanical ventilation, hoping to find out the different manifestations of patients through the investigation by a variety of physiologic measurements, so as to understand whether different types of patients phenotype to derive different clinical strategies for liberation of the mechanical ventilator.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 10 days of mechanical ventilation at the intensive care unit of National Taiwan University Hospital and transferred to the Respiratory Care Center of National Taiwan University Hospital for weaning training
* Patients who have undergone tracheostomy and still have a tracheotomy tube
* Are at least 20 years old
* Stable respiratory condition with inspired oxygen fraction not exceeding 50%

Exclusion Criteria:

* Hemodynamic instability or continuous use of vasopressors
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic critically ill patients receiving prolonged mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2022-07-31 (Actual); Primary Completion 2025-02-17 (Estimated); Study Completion 2025-02-17 (Estimated)

PRIMARY OUTCOMES:
Liberation from mechanical ventilation at discharge from the weaning unit | Five days
  At least five consecutive days of free from mechanical ventilation ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Jih-Shuin Jerng, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan